CLINICAL TRIAL: NCT00368407
Title: Optimal Treatment Frequency of 308-Nm Excimer Laser for Vitiligo on the Face and Neck
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Other Study IDs: fmmu200504
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2005-04

CONDITIONS: Vitiligo
Keywords: 308-nm excimer laser; vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Lasers, Excimer

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: 308-nm excimer laser

SUMMARY:
To determine the optimal treatment frequency of 308-nm excimer laser for vitiligo and identify the key clinical variable(s) associated with the treatment efficiency under the optimal treatment frequency.

Prospective, randomized, comparative study among groups of vitiligo patients treated with 308-nm excimer laser, with the limitation of no follow-up.

DETAILED DESCRIPTION:
Vitiligo patients were treated with 308-nm excimer laser for 20 sessions at different frequencies (0.5×, 1.0×, 2.0× and 3.0× weekly). Treatment protocols adapted the dose to the lesions and not to the minimal erythemal dose. Treatment efficacy was blindly evaluated by 2 independent physicians. Re-pigmentation rate was graded on a 6-point scale. The onset of re-pigmentation of vitiligo lesions was evaluated after 5 treatment sessions. The differences between Group 0.5×, 1.0×, 2.0× and 3.0× linking different clinical variables were assessed.

ELIGIBILITY:
Inclusion Criteria:

* older than 2 years, stable vitiliginous patches during the past 3 months with surfaces of at least 4cm2, and an understanding of all information given by signing a written consent form.

Exclusion Criteria:

* pregnant or breastfeeding women; personal history of a hypertrophic scar, skin cancer; taking immunosuppressive or photosensitizing drugs and undergoing phototherapy during the past 3 months.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2005-04; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: gao tianwen, MD,PHD, Study Director — Ddepartment of Dermatology
Locations (1):
- Department of dermatology, Xijing Hospital, Xi'an, Shannxi, China

REFERENCES:
- [Result] Hofer A, Hassan AS, Legat FJ, Kerl H, Wolf P. Optimal weekly frequency of 308-nm excimer laser treatment in vitiligo patients. Br J Dermatol. 2005 May;152(5):981-5. doi: 10.1111/j.1365-2133.2004.06321.x. PMID 15888156